CLINICAL TRIAL: NCT03050463
Title: Impact of Affect Reactivity and Regulation on Breast Cancer Treatment Decisions
Brief Title: Functional Magnetic Resonance Imaging in Assessing Affect Reactivity and Regulation in Patients With Stage 0-III Breast Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-34959; NCI-2016-01547 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRSADJ0030 (Other: OnCore); U01CA197282 (NIH)
Record Dates: First submitted 2016-11-07; First posted 2017-02-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Healthy Subject; Stage 0 Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- breast cancer with bilateral mastectomy: This group has patients with breast cancer who have chosen to have a bilateral mastectomy. Patients complete questionnaires over 1 hour, undergo fMRI related tasks over 2-2.5 hours, and blood/saliva sample collection upon awakening, 30 minutes after awakening, and at 9 pm in the evening for 3 consecutive days.
  Interventions: Procedure: Biospecimen Collection; Procedure: Functional Magnetic Resonance Imaging; Other: Questionnaire Administration
- breast cancer without bilateral mastectomy: This group has patients diagnosed with breast cancer who have chosen not to have bilateral mastectomy (e.g. they may have unilateral mastectomy, lumpectomy, radiation, etc. but not bilateral mastectomy). Patients complete questionnaires over 1 hour, undergo fMRI related tasks over 2-2.5 hours, and blood/saliva sample collection upon awakening, 30 minutes after awakening, and at 9 pm in the evening for 3 consecutive days.
  Interventions: Procedure: Biospecimen Collection; Procedure: Functional Magnetic Resonance Imaging; Other: Questionnaire Administration
- healthy subjects: Patients complete questionnaires over 1 hour, undergo fMRI related tasks over 2-2.5 hours, and blood/saliva sample collection upon awakening, 30 minutes after awakening, and at 9 pm in the evening for 3 consecutive days.
  Interventions: Procedure: Biospecimen Collection; Procedure: Functional Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and saliva sample collection
Procedure: Functional Magnetic Resonance Imaging — Undergo fMRI related tasks
  Other Names: fMRI; FUNCTIONAL MRI
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The investigators hope to gain a better understanding of the influence of affect reactivity and regulation on the decision of newly diagnosed breast cancer patients to choose bilateral mastectomy. The information gained can help develop an intervention to enable management of cancer-related anxiety by non-surgical means.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine affect reactivity and regulation among women with a recent diagnosis of breast cancer in comparison to healthy controls.

II. Relate affect reactivity and regulation to choice of bilateral mastectomy (BLM).

SECONDARY OBJECTIVES:

I. Assess long term functioning correlates of BLM decision and affect reactivity and regulation.

OUTLINE: Study plans to recruit total of 170 women. Participants will be assigned to 3 arms. For women diagnosed with breast cancer (total of 130) 65 with BLM as part of their cancer treatment and 65 non-BLM. The 3rd arm being 40 women with no cancer diagnosis as controls.

Study protocol will be the same for all 170 Study participants. Active participation by each participant will be approximately 8 hours at baseline and 2 hours at 6, 12, and 18-month follow-ups. Baseline assessment involve completing a set of questionnaires, participating in various tasks while undergoing an MRI scan of the head, providing saliva samples and I tube of blood. Follow-up assessments involve completing a set of questionnaires and saliva collection, all can be done at home.

ELIGIBILITY:
Inclusion Criteria:

Women Diagnosed with breast cancer

* Female
* Age 18 or older
* Agree to suspend treatments containing Benzodiazepines and steroids up to 2 weeks pre and during cortisol sampling (based on PI's clinical judgement)
* Agree to taking saliva samples and having fMRI scan
* No contraindications to MRI imaging (like ferromagnetic metal in their body)
* Proficiency in English sufficient to complete questionnaires and follow instructions during the fMRI assessments
* US Citizen or resident able to receive payment legally
* Documented stage 0-III breast cancer
* Unilateral breast tumors

Controls

* Female
* Age 18 or older
* Agree to suspend treatments containing Benzodiazepines and steroids up to 2 weeks pre and during cortisol sampling (based on PI's clinical judgement)
* Agree to having saliva samples and fMRI scan
* No contraindications to MRI imaging (like ferromagnetic metal in their body)
* Proficiency in English sufficient to complete questionnaires and follow instructions during the fMRI assessments
* US Citizen or resident able to receive payment legally

Exclusion Criteria:

Women Diagnosed with breast cancer

* Other active cancers within the past 10 years other than squamous cell carcinoma of the skin
* Pregnant
* Any significant neurologic disease, such as dementia, multi-infarct dementia, Parkinson's or Huntington's disease, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, stroke, or traumatic brain injury
* Hearing impaired
* Current untreated psychosis, or bipolar disorder, or substance/alcohol abuse/dependence
* Current use of psychotropic (based on PI's clinical judgement) medication 5 or more days a week

Controls

* Cancer diagnosis, current or past
* Pregnant
* Any significant neurologic disease, such as dementia, multi-infarct dementia, Parkinson's or Huntington's disease, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, stroke, or traumatic brain injury
* Hearing impaired
* Current untreated psychosis, or bipolar disorder, or substance/alcohol abuse/dependence
* Current use of psychotropic (based on PI's clinical judgement) medication 5 or more days a week
* Breast cancer diagnosis in 1 first degree relative or 2 or more second degree relatives
* Ovarian cancer diagnosis in 1 first or second degree relative

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with stage 0-III breast cancer at Stanford Cancer Center, as well as healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Explicit Affect Reactivity and Regulation Measured Using functional MRI (fMRI) Reactivity Probes | Up to 18 months
  Multivariate regression analysis will be used to examine affect reactivity among women with a recent diagnosis of breast cancer in comparison to healthy controls at baseline. Functional data will be collected on the explicit affect regulation task (20 minutes) and explicit cancer related affect regulation task (8 minutes). Affect reactivity and cancer-related affect reactivity will be defined by WATCH negative minus WATCH neutral and by WATCH cancer-related negative and WATCH neutral contrast. The larger this value, the greater the affect reactivity. Explicit affect regulation will defined by WATCH negative minus REAPPRAISE negative, and by WATCH negative minus REAPPRAISE cancer-related negative contrasts. The greater this value, the less successful explicit regulation is.
Implicit Affect Reactivity and Regulation Measured Using fMRI Reactivity Probes | Up to 18 months
  Multivariate regression analysis will be used to examine affect reactivity among women with a recent diagnosis of breast cancer in comparison to healthy controls at baseline. Functional data will be collected on the implicit affect regulation task (13 minutes) and implicit cancer-related affect regulation task (13 minutes). Affect reactivity and cancer-related affect reactivity will be defined by incongruent minus congruent trials and incongruent cancer minus congruent cancer-related trials. The greater this value, the more affect reactivity there is. Implicit affect regulation for general affective content will be calculated by post-congruent incongruent trials minus post-incongruent incongruent trials. Similarly, implicit affect regulation for cancer related content will be calculated from the post-congruent incongruent trials minus post-incongruent incongruent trials in the cancer-related adaptation of the task. The greater this value, the less successful implicit regulation is.

SECONDARY OUTCOMES:
Diurnal Slope of Cortisol | Up to 18 months
  Affect management is associated with the diurnal slope of cortisol. The stress of a breast cancer diagnosis and subsequent treatment choices is bound to affect hormonal stress response systems, such as the hypothalamic-pituitary-adrenal axis (HPA). Cortisol levels, measured reliably in saliva, are a meaningful and accessible way of assessing physiological stress response. Salient to this study of affect regulation, the investigators have found that flatter diurnal cortisol slope is associated with higher repressive-defensiveness and less sustained expression of primary negative affect in a group setting.
BLM decision and affective distress | Up to 18 months
  Longitudinal trajectories of affective distress are examined. For this, The Contralateral Prophylactic Mastectomy (CPM) survey consists of 23 items related to decision making, knowledge, risk perceptions, and worry about breast cancer. It was developed based on expert knowledge measuring decision making, risk perceptions, and knowledge outcomes in patients with breast cancer. It showed in a recent study that choice of CPM is related to significant anxiety about cancer coupled with overestimation of the risk of recurrence and therefore of the benefit of the procedure. This will be used to study the link between affect reactivity and regulation and cognitive distortion about risks and benefits.
Functional status as a predictor of longitudinal progression | Up to 18 months
  Functional status is assessed through self-report measures. The "Ways of Coping Checklist" was developed to assess eight fundamental dimensions of the coping process: confrontation, distancing, self-control, seeking social support, accepting responsibility, escape/avoidance, planful problem solving, and positive reappraisal. These dimensions measure two general functions of coping, problem-focused coping and emotion-focused coping. Problem-focused coping is aimed at doing something to change the stressful situation for the better, whereas emotion- focused coping is aimed at regulating emotional distress

OTHER OUTCOMES:
Choice of BLM and reliance on information from nonmedical sources assessed using the Rosenberg questionnaire | Up to 18 months
  As an exploratory analysis, using logistic regression analysis, an examination of whether women who choose BLM report more reliance on information from nonmedical sources such as media and the internet than on medical professionals and family/friends (Rosenberg Questionnaire (29), question 23) will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

REFERENCES:
- [Derived] Zhang JX, Kurian AW, Jo B, Nouriani B, Neri E, Gross JJ, Spiegel D. Emotion regulation and choice of bilateral mastectomy for the treatment of unilateral breast cancer. Cancer Med. 2023 Jun;12(11):12837-12846. doi: 10.1002/cam4.5963. Epub 2023 Apr 21. PMID 37083300

DOCUMENTS (1):
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03050463/ICF_000.pdf